CLINICAL TRIAL: NCT00247494
Title: Effects of Mycophenolate Mofetil (MMF) on Surrogate Markers for Cardiovascular Disease in HIV-1 Infected Patients
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: Myocardh
Record Dates: First submitted 2005-11-01; First posted 2005-11-02 (Estimated); Last update posted 2009-07-22 (Estimated); Status verified 2005-11

CONDITIONS: HIV Infection; Atherosclerosis
Keywords: HIV-1; atherosclerosis; immunomodulation
MeSH Terms: conditions — HIV Infections; Atherosclerosis | interventions — Mycophenolic Acid; BID protein, human

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: mycophenol mofetil (MMF, Cellcept®) 500 mg BID

SUMMARY:
This study is a substudy of the MAN2 -study (Mycophenol mofetil in Antiretroviral Naïve patients 2, see elsewhere in the ClinicalTrials.gov database). In the MAN2 study, HIV-1 infected patients who are not treated with antiretroviral treatment will be randomized to treatment with Mycophenol mofetil (MMF)500 mg BID or a control group without treatment (open label). Both patients randomized to treatment with MMF and patients randomized to the control group will be asked to participate also in this substudy.

In this substudy we want to show whether monotherapy with Mycophenol mofetil (MMF) in patients infected with HIV-1 can reduce acceleration of atherogenesis by attenuating various inflammatory pathways normally involved in progression of atherosclerosis.

DETAILED DESCRIPTION:
* background Immune activation plays an important role in atherogenesis. In HIV-1 infection, the immune system is chronically hyperactivated. There also seems to be an increased incidence of cardiovascular disease in untreated HIV-1 infection. Mycophenol mofetil (MMF) will be used to treat this immune activation in untreated HIV-1 infected patients in the MAN2-study (see elsewhere in this ClinicalTrials.gov database).
* Hypothesis T-cell inhibition with MMF attenuates T-cell number, T-cell activation and T-cell - monocyte interaction, thereby minimizing the T-cell-driven inflammatory amplification loop.

In addition, MMF reduces expression of adhesion molecules on endothelial cells and leucocytes, thereby attenuating recruitment of circulating leucocytes to the atherosclerotic plaque. Combining these effects MMF treatment will improve anti-atherogenic defence mechanisms, such as improvement of endothelial function and attenuation of the pro-inflammatory state.

*design This will be a substudy of of the multi-center, double-blind, randomized, trial "Mycophenol mofetil in Antiretroviral Naïve patients 2 (MAN2 study)" (called the main study hereafter). The aim of the substudy is to evaluate the effects of mycophenolate mofetil on ´surrogate markers´ for atherosclerosis in a group of HIV-1 infected patients. All 90 patients to be included in the main study will be asked to participate in this substudy. A separate informed consent is needed.

Patients participating in this substudy will undergo study procedures for the substudy only on day 0 and week 48 of the main study (i.e. before the first dose of MMF and after 48 weeks of MMF treatment for the patients randomized to MMF treatment). Extra blood will be drawn to measure several biochemical markers associated with atherosclerosis and will be measured. Furthermore measurements of the condition of the blood vessels will be performed (using ultrasound, amongst others).

ELIGIBILITY:
Inclusion Criteria:

* Any patient included in the MAN2-study van enter this substudy (see protocol MAN2 study)

Exclusion Criteria:

* Any condition, illness or use of medication which according to the investigator is not compatible with the conduct of the substudy or which could interfere with the evaluations required by the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2005-04

PRIMARY OUTCOMES:
The difference between the two groups (patients treated with MMF and the control group without treatment) in the change (week 0-week 48) in biochemical markers, Flow Mediated Dilation and Intima Media Thickness.

SECONDARY OUTCOMES:
The change (week 0-week 48) within patients in biochemical markers, Flow Mediated Dilation and Intima Media Thickness.

CONTACTS AND LOCATIONS:
Overall Officials: Erik S Stroes, MD PhD, Principal Investigator — Department of Internal Medicine, Division of Vascular Medicine, Academic Medical Center, University of Amsterdam
Locations (1):
- Department of Internal Medicine, Academic Medical Center, University of Amsterdam, The Netherlands, Amsterdam, North Holland, Netherlands

REFERENCES:
- [Background] Allison AC, Eugui EM. Mycophenolate mofetil and its mechanisms of action. Immunopharmacology. 2000 May;47(2-3):85-118. doi: 10.1016/s0162-3109(00)00188-0. PMID 10878285
- [Background] Romero F, Rodriguez-Iturbe B, Pons H, Parra G, Quiroz Y, Rincon J, Gonzalez L. Mycophenolate mofetil treatment reduces cholesterol-induced atherosclerosis in the rabbit. Atherosclerosis. 2000 Sep;152(1):127-33. doi: 10.1016/s0021-9150(99)00458-x. PMID 10996347
- [Background] Greenstein SM, Sun S, Calderon TM, Kim DY, Schreiber TC, Schechner RS, Tellis VA, Berman JW. Mycophenolate mofetil treatment reduces atherosclerosis in the cholesterol-fed rabbit. J Surg Res. 2000 Jun 15;91(2):123-9. doi: 10.1006/jsre.2000.5919. PMID 10839960